CLINICAL TRIAL: NCT06616532
Title: A Multicenter, Open-lable, Randomized Phase III Study of PM8002 in Combination With Paclitaxel Compared With Chemotherapy as Second-line Treatment in Small Cell Lung Cancer
Brief Title: PM8002 in Combination With Paclitaxel Compared With Chemotherapy as Second-line Treatment in Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-C014C-SCLC-R
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: SCLC
Keywords: Second-line
MeSH Terms: interventions — Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PM8002+Paclitaxel (Experimental): Subjects will be administered with PM8002 in combination with Paclitaxel via intravenously (IV) infusion.
  Interventions: Drug: PM8002; Drug: Paclitaxel
- Chemotherapy (Active Comparator): Subjects will be administered with Investigator's Choice(Topotecan or Paclitaxel) via intravenously (IV) infusion Q3W.
  Interventions: Drug: Paclitaxel; Drug: Topotecan

INTERVENTIONS:
Drug: PM8002 — Following a predefined dose and date.
  Arms: PM8002+Paclitaxel
Drug: Paclitaxel — 175mg/m2 via IV infusion on Day 1 Q3W
Drug: Topotecan — 1.25mg/m2/day via IV infusion on Days 1-5 Q3W
  Arms: Chemotherapy

SUMMARY:
PM8002 is a bispecific antibody targeting PD-L1 and VEGF. This study will evaluate the efficacy and safety of PM8002 in combination with Paclitaxel as second-line treatment for SCLC

DETAILED DESCRIPTION:
This multicenter, randomized, open-label phase III study will evaluate the efficacy and safety of PM8002 in combination with Paclitaxel versus Investigator's Choice (Topotecan or Paclitaxel) as second-line treatment for subjects with SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this clinical study; full understanding of the study and voluntary signing the informed consent form; willing to follow and abling to complete all trial procedures;
2. Age ≥18 years but ≤75 years;
3. Histologically or cytologically confirmed SCLC;
4. Advanced SCLC that has progressed or replased after first-line platinum-containing chemotherapy (extensive-stage patients must have received immune checkpoint inhibitors);
5. Having adequate organ functions;
6. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;
7. Life expectancy of 12 weeks or more;
8. Having at least one measurable tumor lesion according to RECIST v1.1;

Exclusion Criteria:

1. History of severe allergic disease, severe drug allergy or have known allergy to any component of the study drugs;
2. Previous treatment with Paclitaxel or Topotecan or anti-vascular endothelial growth factor (VEGF) target drugs;
3. Current presence of severe superior vena cava syndrome and spinal cord compression;
4. Adverse events resulting from prior anti-tumor therapies should be assessed and graded according to the CTCAE 5.0 criteria, subjects whose AEs have not returned to Grade 1 or below;
5. Evidence of significant clotting disorder or other significant bleeding risk;
6. History of severe, uncontrollable, or active cardiovascular diseases within 6 months;
7. Current presence of uncontrollable pleural, pericardial, and peritoneal effusions;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome;
9. History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
10. History of alcohol abuse, psychotropic substance abuse or drug abuse;
11. Pregnant or lactating women;
12. Other conditions considered unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 32 months from first patient in
  Overall survival is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis are censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) assessed by evaluated by investigator | Up to approximately 32 months from first patient in
  PFS is defined as the time from randomization to the first documented PD per RECIST 1.1 based on assessments by investigator or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Objective response rate (ORR) evaluated by investigator | Up to approximately 32 months from first patient in
  ORR is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experienced a CR or PR as assessed by investigators based on RECIST 1.1 is presented.
Disease control rate (DCR) | Up to approximately 32 months from first patient in
  DCR is defined as the sum rate of CR, PR and Stable Disease (SD), as determined by investigators based on RECIST v1.1
Time to response (TTR) | Up to approximately 32 months from first patient in
  Time to response(TTR) is defined as the time from randomization to the first documented PR or CR assssed by investigator based on RECIST v1.1
Duration of response (DOR) | Up to approximately 32 months from first patient in
  DoR is defined as the time period from the date of initial CR or PR until the date of PD or death due to any cause, whichever occurs first.
6 month PFS rate | Up to approximately 32 months from first patient in
  PFS rate corresponding to the 6th month of the progression-free survival curve
12 month PFS rate | Up to approximately 32 months from first patient in
  PFS rate corresponding to the 12th month of the progression-free survival curve
12 month OS rate | Up to approximately 32 months from first patient in
  OS rate corresponding to the 12th month of the overall survival curve
Incidence and severity of Adverse Event (AE) according to CTCAE 5.0 | Up to 30 days after last treatment
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  To evaluate the incidence and characteristics of ADA to PM8002
Health related quality of life (HRQoL) | Up to 30 days after last treatment
  Differences in the scores of health-related quality of life (HRQol)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (45):
- China (45):
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital Of Ningbo University, Ningbo, Zhejiang
  - Binzhou Medical University Hospital, Binzhou
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - First People's Hospital of Chenzhou, Chenzhou
  - The First Affiliated Hospital of Army Medical University, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - The First People's Hospital of Foshan, Foshan
  - Fujian Cancer Hospital, Fuzhou
  - The Affiliated Hospital Of Guilin Medical University, Guilin
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Hospital, Hefei
  - Shandong Cancer Institute, Jinan
  - Jingzhou First People's Hospital, Jingzhou
  - Affiliated Hospital of Jining Medical University, Jining
  - Yunnan Cancer Hospital, Kunming
  - Liuzhou People's Hospital, Liuchow
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang
  - Meizhou People's Hospital, Meizhou
  - Mianyang Central Hospital, Mianyang
  - Jiangxi Cancer Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanchong Central Hospital, Nanchong
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum-Tower Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Nanyang Central Hospital, Nanyang
  - Qujing NO.1 Hospital, Qujing
  - The Fourth Hospital of Hebei Medical University, Shijia Zhuang
  - Taizhou Enze Medical Center (group), Taizhou
  - Weifang NO.2 People's Hospital, Weifang
  - Weihai Municipal Hospital, Weihai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital Of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - Xuzhou Central Hospital, Xuzhou
  - The Second People's Hospital Of Yibin, Yibin
  - Yongzhou Central Hospital, Yongzhou
  - Yuncheng City Center Hospital, Yuncheng
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou
  - Zhoukou Central Hospital, Zhoukou

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations.
Time Frame: After the trial completed.
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.